CLINICAL TRIAL: NCT01758380
Title: A Double Blind, Double Dummy, Randomised, Multi-centre Study to Assess the Tolerability and Efficacy Profile of Vildagliptin Compared to Gliclazide as Dual Therapy With Metformin in Muslim Patients With Type 2 Diabetes Fasting During Ramadan
Brief Title: Vildagliptin Compared to Gliclazide as Dual Therapy With Metformin in Muslim Patients With Type 2 Diabetes Fasting During Ramadan
Acronym: STEADFAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A2411; 2011-005499-41 (EudraCT Number)
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Ramadan; Vildagliptin; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Vildagliptin; Gliclazide; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin + placebo to Gliclazide (Experimental): Vildagliptin tablets will be given at 50mg twice daily (bid). Placebo to Gliclazide capsules will be given at an equivalent dose to previous sulfonylurea in multiples of 80mg only (80-320 mg/day). Patients will continue their open-label metformin therapy at dosage between 1500-2500 mg daily.
  Interventions: Drug: Vildagliptin; Drug: Metformin; Drug: Placebo to Gliclazide
- Gliclazide + placebo to Vildagliptin (Active Comparator): Gliclazide capsules will be given in multiples of 80 mg (80-320 mg/day) at a dose equivalent to previous sulfonylurea dose, unless at the investigator's discretion it could be up-titrated to the next available dose (if HbA1c is higher than 7.5%). Placebo to Vildagliptin tablets will be given at 50mg twice daily (bid). Patients will continue their open-label metformin therapy at dosage between 1500-2500 mg daily.
  Interventions: Drug: Gliclazide; Drug: Metformin; Drug: Placebo to Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Patients will be instructed to take Vildagliptin tablets at a fixed dose of 50 mg twice daily (double blind therapy)
  Other Names: Galvus
  Arms: Vildagliptin + placebo to Gliclazide
Drug: Gliclazide — Patients will be instructed to take Gliclazide capsules at an equivalent dose to previous sulfonylurea in multiples of 80mg only (double blind therapy)
  Arms: Gliclazide + placebo to Vildagliptin
Drug: Metformin — Patients in both arms will take Metformin at a dose between 1500mg-2500mg per day, in an open label fashion
Drug: Placebo to Gliclazide — Patients will be instructed to take the Gliclazide matching placebo capsules at an equivalent dose to previous sulfonylurea in multiples of 80mg only (double blind therapy)
  Arms: Vildagliptin + placebo to Gliclazide
Drug: Placebo to Vildagliptin — Patients will be instructed to take Vildagliptin matching placebo tablets at a fixed dose of 50 mg twice daily (double blind therapy).
  Arms: Gliclazide + placebo to Vildagliptin

SUMMARY:
To evaluate vildagliptin as compared to gliclazide, given in combination with metformin in Muslim patients with type 2 diabetes fasting during Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Type 2 Diabetes diagnosis
* Plan to fast during Ramadan
* Treated with a combination of metformin and an Sulfonylurea (SU) for at least 12 weeks and HbA1c ≤8.5% at Visit 1
* Taking a sulfonylurea treatment for less than 3 years prior to Visit 1
* Body mass index (BMI) ≥22 and ≤45 kg/m2 at Visit 1

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
* Patients who are taking any other anti-diabetes drug (oral or injection) other than metformin and an SU component.
* Inability to comply with the study procedures or medications.

"Other protocol-defined inclusion/exclusion criteria may apply"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients experiencing at least one Hypoglycaemic Event (HE) during the Ramadan fasting period to test superiority | 1 month

SECONDARY OUTCOMES:
Percentage of patients without an increase in HbA1c (≤ 0.3%) and with no Hypoglycaemic Events (HEs) | visit 3 (anytime from week -4 to day -1 before start of Ramadan) to visit 4 (within 4 weeks post-Ramadan fasting period) (minimum 4.5 weeks to maximum 12 weeks) for HbA1c; and during 1 month (Ramadan) for HEs
Change from baseline to endpoint in glycosylated hemoglobin (HbA1c) | baseline to visit 4 (within 4 weeks post-Ramadan fasting period) (minimum 12.5 weeks to maximum 30 weeks)
  Endpoint is defined as the visit 4 (post-Ramadan) measurement or the last observation obtained during or after Ramadan, prior to or at initiation of rescue medication
Change from visit 3 (pre-Ramadan visit) to endpoint in glycosylated hemoglobin (HbA1c) | visit 3 (anytime from week-4 to day-1 before start of Ramadan) to visit 4 (within 4 weeks post-Ramadan fasting period) (minimum 4.5 weeks to maximum 12 weeks)
  Endpoint is defined as the visit 4 (post-Ramadan) measurement or the last observation obtained during or after Ramadan, prior to or at initiation of rescue medication
Proportion of patients experiencing severe hypoglycemic events during the Ramadan fasting period | 1 month
mean amplitude of glycemic excursions (MAGE) to measure glucose fluctuations during the day | 72 hours
  assessed in a selected subgroup of patients
Treatment adherence during the Ramadan fasting period | 1 month
Change from visit 3 (pre-Ramadan visit) to endpoint in body weight | From visit 3 (anytime from week-4 to day-1 before start of Ramadan) to visit 4 (within 4 weeks post-Ramadan fasting period) (minimum 4.5 weeks to maximum 12 weeks)
  Endpoint is defined as the visit 4 (post-Ramadan) measurement or the last observation obtained during or after Ramadan, prior to or at initiation of rescue medication
Number of unscheduled visit to health care professional | From visit 3 (anytime from week-4 to day-1 before start of Ramadan) to visit 4 (within 4 weeks post-Ramadan fasting period) (minimum 4.5 weeks to maximum 12 weeks)
Number of days fasted during the Ramadan fasting period | 1 month
Number of patients with treatment emergent adverse events (AEs), serious AEs, discontinuation due to AEs, deaths or laboratory abnormalities as assessment of safety and tolerability | Baseline to visit 4 (within 4 weeks post-Ramadan fasting period) (minimum 12.5 weeks to maximum 30 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Director — Novartis Pharmaceuticals
Locations (58):
- Novartis Investigative Site, Frederiksberg, Denmark
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- Germany (9):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Einbeck
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Meine
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Saarlouis
- Indonesia (4):
  - Novartis Investigative Site, Malang, East Java
  - Novartis Investigative Site, Surabaya, East Java
  - Novartis Investigative Site, Jakarta, Jakarta Special Capital Region
  - Novartis Investigative Site, Padang, West Sumatra
- Novartis Investigative Site, Amman, Amman Governorate, Jordan
- Novartis Investigative Site, Kuwait City, Kuwait, Kuwait
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Hazmiyeh
  - Novartis Investigative Site, Saida
- Malaysia (2):
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Kuala Lumpur
- Russia (6):
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Ufa
- Saudi Arabia (2):
  - Novartis Investigative Site, Dammam, Dammam
  - Novartis Investigative Site, Riyadh
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Spain (8):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, Salt, Catalonia
  - Novartis Investigative Site, Santa Coloma de Gramanet, Catalonia
  - Novartis Investigative Site, Vic, Catalonia
  - Novartis Investigative Site, Ceuta, Ceuta
  - Novartis Investigative Site, Melilla, Melilla
- Tunisia (6):
  - Novartis Investigative Site, Monastir, Tunisia
  - Novartis Investigative Site, Le Belvedere - Tunis, Tunisie
  - Novartis Investigative Site, Sfax, Tunisie
  - Novartis Investigative Site, Tunis, Tunisie
  - Novartis Investigative Site, Sousse
  - Novartis Investigative Site, Tunis
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Diskapi / Ankara, Turkey
  - Novartis Investigative Site, Istanbul, Turkey
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kahramanmaraş
- Novartis Investigative Site, Dubai, United Arab Emirates
- United Kingdom (6):
  - Novartis Investigative Site, Leicester, Leicestershire
  - Novartis Investigative Site, London, London
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bolton
  - Novartis Investigative Site, Derby
  - Novartis Investigative Site, Manchester

REFERENCES:
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938
- [Derived] Hassanein M, Abdallah K, Schweizer A. A double-blind, randomized trial, including frequent patient-physician contacts and Ramadan-focused advice, assessing vildagliptin and gliclazide in patients with type 2 diabetes fasting during Ramadan: the STEADFAST study. Vasc Health Risk Manag. 2014 May 28;10:319-26. doi: 10.2147/VHRM.S64038. eCollection 2014. PMID 24920915